CLINICAL TRIAL: NCT04851548
Title: Evaluate the Effectiveness of Bioactive Hyaluronic Acid in the Treatment of Furcation Involvement
Brief Title: Evaluate the Effect of Hyaluronic Acid in the Treatment of Furcation Involvement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Riyadh Elm University (Other)
Responsible Party: Principal Investigator, Ghady Adnan Alqahtani, periodontic resident, Riyadh Elm University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FPFGRP/2021/566
Record Dates: First submitted 2021-03-03; First posted 2021-04-20 (Actual); Last update posted 2021-09-17 (Actual); Status verified 2021-09

CONDITIONS: Furcation Defects
Keywords: Hyaluronic Acid; Furcation involvement
MeSH Terms: conditions — Furcation Defects | interventions — Hyaluronic Acid

STUDY DESIGN:
Intervention Model Description: test group use membrane and hyaluronic acid ,control group use membrane without hyaluronic acid
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (control) (Active Comparator): preoperative cone-beam computed tomography (CBCT) scans N=9
  * open flap debridement.
  * use membrane without hyaluronic acid. (The first monitor will be done after three months. The data will be recorded. After another three months, the patients will undergo an x-ray check again, and the data will be registered. The goal is to have the patients exposed to x-ray twice not to be compromised to a high radiation dose. The evaluation to be done for the 3-month interval will only be clinical assessments|)
  Interventions: Procedure: hyaluronic acid
- Group B (test) (Active Comparator): preoperative cone-beam computed tomography (CBCT )scans N= 9
  * open flap debridement.
  * use membrane and 8% hyaluronic acid gel (The first monitor will be done after three months. The data will be recorded. After another three months, the patients will undergo an x-ray check again, and the data will be registered. The goal is to have the patients exposed to x-ray twice not to be compromised to a high radiation dose. The evaluation to be done for the 3-month interval will only be clinical assessments|).
  Interventions: Procedure: hyaluronic acid

INTERVENTIONS:
Procedure: hyaluronic acid — after flap refection, the furcation area will be debrided then add hyaluronic acid 8% and cover it with a collagen membrane

SUMMARY:
the effect Hyaluronic Acid in the Treatment of Furcation Involvement

DETAILED DESCRIPTION:
The materials to be used in the study are the following:

* Hyaluronic acid
* Cone-beam computed tomography(CBCT) x-ray The patients with Grade II furcation will be divided into two groups. Both groups will have the same number of patients and the same procedure, such as the scaling root planning. However, the control group will use hyaluronic acid and membrane. The placebo group, on the other hand, will use hyaluronic acid without membrane and will use CBCT x-ray. The x-rays will be done at the beginning of the treatment. Then, two monitoring processes will be done. The first monitor will be done after three months. The data will be recorded. Then, after another three months, the patients will undergo an x-ray check again, and the data will be recorded. The goal is only to have the patients exposed to x-ray twice so they would not be compromised to the high dose of radiation. The evaluation to be done for the 3-month interval will only be clinical assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Selected teeth: Permanent first and second molars in the mandible.
2. Furcation dimension: Radiographic and clinical evidence of exhibiting defects due to Grade II furcation with at least 2 millimeters probing depth horizontally and at least 5 millimeters probing depth circumferential.
3. Gender: both males and females.
4. Age range: between 18 and 55 years.
5. Health status: healthy patients non-systemic diseased except controlled diabetic.
6. Compliance: Patients will be willing and able to comply with adequate oral hygiene protocols.

Exclusion Criteria:

1. Patients that received periodontal regenerative therapy within the past 12 months.
2. Patients that are lactating.
3. Pregnant patients.
4. Smokers.
5. Patients with pulp infection.
6. Patients with trauma resulting from occlusion.
7. Patients with receding gum.
8. Patients with tooth mobility greater than grade II.
9. Patients that will not comply with the hygiene protocols in Phase I therapy.
10. Patients with potential illnesses that can influence the periodontal therapy outcomes.
11. Patients that are taking medications that can interfere with the healing outcomes of the periodontal wound.
12. Patients allergic to any drugs.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Estimated)
Dates: Start 2021-09-23 (Estimated); Primary Completion 2022-09-20 (Estimated); Study Completion 2022-09-20 (Estimated)

PRIMARY OUTCOMES:
evaluate the regenerative effect of hyaluronic acid | 6 months
  measurement of the bone gain after the treatment with hyaluronic acid in millimeters

CONTACTS AND LOCATIONS:
Overall Officials: ahmed t gamal, clinical MD, Study Director — Riyadh Elm University

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Kalra SH, Monga C, Kalra KH, Kalra SH. A roentgenographic assessment of regenerative efficacy of bioactive Gengigel((R)) in conjunction with amnion membrane in grade II furcation defect. Contemp Clin Dent. 2015 Apr-Jun;6(2):277-80. doi: 10.4103/0976-237X.156068. PMID 26097373
- [Background] Sahayata VN, Bhavsar NV, Brahmbhatt NA. An evaluation of 0.2% hyaluronic acid gel (Gengigel (R)) in the treatment of gingivitis: a clinical & microbiological study. Oral Health Dent Manag. 2014 Sep;13(3):779-85. PMID 25284557
- [Result] Ainamo J, Bay I. Problems and proposals for recording gingivitis and plaque. Int Dent J. 1975 Dec;25(4):229-35. PMID 1058834
- [Result] Gaurav Bakutra., et al. "Prevalence, Extension and Severity Associated Risk Factors Associated with Furcation Involvement in an Adult Population. An Epidemiological Study
- [Result] Bjorn H, Halling A, Thyberg H. Radiographic assessment of marginal bone loss. Odontol Revy. 1969;20(2):165-79. No abstract available. PMID 5259016
- [Result] Carranza, F. A. & Newman, M. G., 2018. Clinical Periodontology. USA: WB Saunders & Co.
- [Result] Glickman, I. (1972). Clinical Periodontology: Prevention, Diagnosis, and Treatment of Periodontal Disease in the Practice of General Dentistry (4th ed.). Saunder.
- [Result] Pilloni A, Rojas MA. Furcation Involvement Classification: A Comprehensive Review and a New System Proposal. Dent J (Basel). 2018 Jul 23;6(3):34. doi: 10.3390/dj6030034. PMID 30041399
- [Result] Sandhu GK, Khinda PK, Gill AS, Kalra HS. Surgical re-entry evaluation of regenerative efficacy of bioactive Gengigel((R)) and platelet-rich fibrin in the treatment of grade II furcation: A novel approach. Contemp Clin Dent. 2015 Oct-Dec;6(4):570-3. doi: 10.4103/0976-237X.169855. PMID 26681869
- [Result] Sakpal TV. Sample size estimation in clinical trial. Perspect Clin Res. 2010 Apr;1(2):67-9. PMID 21829786
- [Result] https://doi.org/10.1902/jop.1959.30.1.7